CLINICAL TRIAL: NCT02897505
Title: Evaluating the Effect of Music on Emotional Regulation Among Survivors of Sexual Violence
Brief Title: Music Workshops in the EMPOWER Clinic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling subjects
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-01524
Record Dates: First submitted 2016-08-30; First posted 2016-09-13 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Sex Trafficking; Sexual Violence; Trauma
Keywords: post traumatic stress disorder (PTSD)
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Women enrolled in Empower Clinic (Experimental): Women who are enrolled in the Empower Sanctuary will be asked to participate in a Music Workshop
  Interventions: Behavioral: Music Workshop

INTERVENTIONS:
Behavioral: Music Workshop — At each music workshop, the study staff will collect participants' pre- and post-session Physiological and Emotional Thermometer Surveys. The pre-session survey will be conducted prior to the start of the music workshop, and the post-session survey will be conducted within 15 minutes after the conclusion of the workshop.

SUMMARY:
Women will be recruited from the EMPOWER clinic when they present for care; they may be given a flyer as part of their clinic entry paperwork, or approached by a study staff member in the waiting area of the clinic. Women who are clients of Sanctuary for Families may find out about the music workshops and the study through Sanctuary for Families staff, who will post flyers in their noticeboards or offices.

This study will use a repeated measures survey design to evaluate the effect of a musical workshop intervention to aid in the management of mood, anxiety, and stress among women enrolled in the EMPOWER clinic for survivors of sex trafficking and sexual violence. Assessment of the feasibility and acceptability of this music intervention will be carried out on participants as they are taught to manage stress and emotions.

ELIGIBILITY:
Inclusion Criteria:

* Women enrolled in the EMPOWER clinic and/or Sanctuary for Families

Exclusion Criteria:

* Unwilling or unable to participate or provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety, and Stress Scale (DASS-21) | Baseline to Three (3) Months
  The DASS-21 is a 21-item self-report questionnaire that measures the severity of a range of core depression, anxiety, and stress symptoms. [6] The DASS-21 has been translated and validated in many languages, including Spanish, French and Chinese. In this study, the DASS-21 is conducted three times: at the beginning of the study (pre-intervention), at the end of the study (post-intervention), and at 3 months after the study (3-month follow-up). The DASS-21 can be completed in 5-7 minutes.

SECONDARY OUTCOMES:
Life Events Checklist (LEC-5): | Baseline to Three (3) Months
  The LEC is a widely used self-report questionnaire that assesses participants' exposure to 16 potentially traumatic events and one additional stressful event not captured in the other 16 items. The LEC has been translated and validated in many languages, and can be completed in 5-7 minutes.
Physiological and Emotion Thermometers Survey | Baseline to Three (3) Months
  The Physiological and Emotion Thermometers Survey records information on participants' physiological indicators (heart rate and blood pressure) and self-reported answers on the Emotion Thermometers, which is a simple visual-analogue tool used to detect and monitor emotional disorders and has been translated in many languages including Spanish, French and Chinese. The survey is conducted at the beginning and at the end of each music workshop (pre- and post-session, respectively) that the participant attends, and can be completed in 2-5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Ades, MD, Principal Investigator — New York University Medical School